CLINICAL TRIAL: NCT01398670
Title: Comparison of the Immunogenicity of Wockhardt's Insulin Analogue Lispro and Lispro Mix With Eli Lilly's Insulin Analogue Humalog® and Humalog® Mix in Type 1 Diabetic Patients
Brief Title: Immunogenicity Study of Wockhardt's Insulin Lispro/Lispro Mix Basal Bolus Regimen in Type 1 Diabetics
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not initiated
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P3-LIS-IMSFDA-01
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Type I Diabetes
Keywords: Type I Diabetes; Wockhardt's Insulin analogue Lispro; Humalog®; Humalog Mix; Wockhardt; Biosimilar; Phase 3
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lispro arm (Experimental): Lispro and Lispro Mix 75/25 /Lispro Mix 50/50
  Interventions: Biological: Insulin Lispro
- Humalog® arm (Active Comparator): Humalog® and Humalog® Mix75/25 / Humalog® Mix50/50
  Interventions: Biological: Insulin Lispro

INTERVENTIONS:
Biological: Insulin Lispro — a. Lispro and Lispro Mix® 75/25 / Lispro Mix 50/50
  The drugs would be administered subcutaneously
  Arms: Lispro arm
Biological: Insulin Lispro — Humalog® and Humalog® Mix75/25 /Humalog® Mix 50/50
  The drugs would be administered subcutaneously
  Arms: Humalog® arm

SUMMARY:
This is a randomized, parallel group comparison of the immunogenicity safety of Wockhardt's Insulin analogue Lispro and lispro Mix with Eli Lilly's Insulin analogue Humalog® and Humalog® Mix in patients with Type 1 Diabetes Mellitus

DETAILED DESCRIPTION:
To evaluate and compare the Immunogenicity safety of Wockhardt's Insulin analogue Lispro and lispro Mix with Eli Lilly's Insulin analogue Humalog® and Humalog® Mix in Type I Diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who understand the nature of the study and are willing to provide written informed consent.
2. Patients who have been pre-diagnosed as cases of type-1 diabetes for a period not less than 1 year
3. Male or Female Patients ≥ 18 and < 55 years of age.
4. Patients with body mass index (BMI) of 18.0 to 30.0 kg/m2
5. Patients who are cooperative, reliable, and agree to have regular injections of insulin and are willing to comply with protocol procedures.
6. Ability to use the self glucose-monitoring device and to self inject insulin.

Exclusion Criteria:

1. Females who are pregnant or lactating, or not practicing adequate contraception.
2. A Patient with compromised hepatic or renal function
3. A Patient who is an employee of the Investigator, or a patient who has a direct involvement with the trial or other trials under the direction of the Investigator.
4. A Patient who has been treated with other investigational agent or devices within the previous 30 days, has planned use of investigational drugs or devices, or has been previously randomized in this trial.
5. A Patient with history or evidence of allergy to insulin preparations.
6. A Patients who is currently receiving or has received, within the last year, any immunomodulator medications.
7. Patients unlikely to comply with the study protocol e.g. unable to return periodically for subsequent visits.
8. Patients who are judged by the investigator as inappropriate to participate in the study for any reason other than those mentioned.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months

SECONDARY OUTCOMES:
Percentage change in the immunogenic response | 6 months
Correlation of the immunogenicity with hypoglycemia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Rasendrakumar Jha, Study Director — Wockhardt